CLINICAL TRIAL: NCT04710212
Title: Screening for Colonization With Resistant Enterobacterales in Neutropenic Patients With Hematologic Malignancies (SCENE)
Brief Title: Screening for Colonization With Resistant Enterobacterales in Neutropenic Patients With Hematologic Malignancies
Acronym: SCENE
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Weill Medical College of Cornell University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00106363; UM1AI104681 (NIH)
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Hematologic Malignancy; Leukemia, Acute; Neutropenia; Bloodstream Infection
Keywords: FQRE; Fluoroquinolone-resistant Enterobacterales; Hematopoietic stem cell transplantation; HCT; Induction chemotherapy; Hematologic Malignancy; Acute Leukemia; Neutropenia; Bloodstream infection; Perianal swab; Gram-negative bacteremia
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Neutropenia; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Perianal swabs are collected from subjects and only isolates are retained. Bloodstream infection isolates are retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Induction Chemotherapy for Acute Leukemia: Receiving induction chemotherapy for acute leukemia, and receiving fluoroquinolone (FQ) prophylaxis.
  Interventions: Other: No intervention.
- Hematopoietic stem cell transplantation (HCT): Undergoing hematopoietic stem cell transplantation (HCT), and receiving fluoroquinolone (FQ) prophylaxis.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — Observational study with no intervention.

SUMMARY:
This is a prospective, observational cohort study to assess the frequency with which neutropenic patients with hematologic malignancies and hematopoietic cell transplant (HCT) recipients are colonized with fluoroquinolone-resistant Enterobacterales (FQRE) and the clinical impact of FQRE colonization.

DETAILED DESCRIPTION:
This is a prospective, observational cohort study to assess the frequency with which neutropenic patients with hematologic malignancies and hematopoietic cell transplant (HCT) recipients are colonized with fluoroquinolone-resistant Enterobacterales (FQRE) and the clinical impact of FQRE colonization.

The investigator will collect perianal swabs from patients receiving induction chemotherapy for acute leukemia or undergoing hematopoietic stem cell transplantation (HCT), and who are receiving fluoroquinolone (FQ) prophylaxis. FQRE colonization will be assessed by culture, and the investigator will correlate FQRE colonization with the risk of Gram-negative bacteremia during neutropenia.

Population: 410 adults with acute leukemia who are receiving induction chemotherapy and HCT recipients who are receiving FQ prophylaxis during neutropenia.

Results of this study will be combined with a portion of subject data from an identically-designed R01-funded study of FQRE colonization. The combined data will be used for study analysis and reporting.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent
2. Male or female ≥18 years of age
3. Receiving intensive induction chemotherapy for acute leukemia or undergoing HCT
4. Receive fluoroquinolone prophylaxis during neutropenia

Exclusion Criteria:

1. Expected to have <7 days of neutropenia (absolute neutrophil count ≤500 cells/μL) after receipt of chemotherapy (a) (acute leukemia cohort only)
2. First swab collected ≥5 days after onset of chemotherapy
3. First swab collected after the day of transplant (HCT cohort only)
4. Acute promyelocytic leukemia
5. Receiving chimeric antigen receptor (CAR)-T-cell therapy
6. Pregnant women as determined by clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 410 adults with acute leukemia who are receiving induction chemotherapy and HCT recipients who are receiving FQ prophylaxis during neutropenia.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Gram-negative bloodstream infection (BSI) | Until neutrophil recovery or 30 days after collection of the first swab in patients who do not have neutrophil recovery by 30 days
  Gram-negative BSI during the episode of neutropenia

SECONDARY OUTCOMES:
Colonization with FQRE and ESBL-E | Within 4 days after initiation of chemotherapy
  Colonization with fluoroquinolone-resistant Enterobacterales (FQRE) and Extended-spectrum-beta-lactamase-producing Enterobacterales (ESBL-E) upon initiation of chemotherapy
Fever | Until neutrophil recovery or 30 days after collection of the first swab in patients who do not have neutrophil recovery by 30 days
  Occurrence (Yes/No) of fever (≥38.0°C) during the episode of neutropenia.
Bloodstream infection (BSI) | Until neutrophil recovery or 30 days after collection of the first swab in patients who do not have neutrophil recovery by 30 days
  Any BSI during the episode of neutropenia
Intensive care unit (ICU) admission | Prior to neutrophil recovery or 30 days after collection of the first swab in patients who do not have neutrophil recovery by 30 days
  Intensive care unit admission prior to recovery from neutropenia
90-day mortality | Occurs within 90 days from the collection of the first swab
  90-day mortality from the collection of the first swab

OTHER OUTCOMES:
Incidence of and risk factors for acquiring FQRE and ESBL-E during the episode of neutropenia | During the episode of neutropenia, up to 30 days
  Acquisition of FQRE and ESBL-E in patients not initially colonized with these organisms

CONTACTS AND LOCATIONS:
Overall Officials: Michael Satlin, Principal Investigator — Weill Medical College of Cornell University; Vance G Fowler, MD, Study Director — Duke Clinical Research Institute
Locations (6):
- United States (6):
  - University of California San Fransisco Medical Center, San Francisco, California
  - Hackensack Meridian Health, Nutley, New Jersey
  - Mount Sinai Hospital, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No